CLINICAL TRIAL: NCT07388823
Title: Nail Bed Repair RCT
Brief Title: Nailbed Repair for Patients With Nailbed Injuries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anna Luan, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 82680
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Nail Bed Injury; Nail Place Disruption; Nail Laceration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irrigation and Dressing (Active Comparator): Patients in this arm will receive the following treatment protocol:
  1. If there is a subungual hematoma >50% of the nail, trephinate the nail plate using an 18G needle
  2. Irrigate wound with at least 500cc normal saline
  3. Dress finger with bacitracin, xeroform, and 2" kling wrap
  4. Splint finger as needed with alumifoam splint (apply splint to volar side of finger so as to avoid pressure to nail bed)
  5. Repair any other lacerations as needed
  Interventions: Other: Nail bed dressing
- Nail bed repair (Experimental): Patients in this arm will receive the following treatment protocol:
  1. Block involved digit with 3cc 1% lidocaine injected subcutaneously over volar and dorsal metacarpophalangeal joint
  2. Apply tourniquet to base of finger if desired
  3. Remove nail using freer/hemostats
  4. Irrigate wound with at least 500cc normal saline
  5. Repair nail bed laceration with 5-0 chromic or monocryl suture
  6. Stent eponychium with native nail or fashion substitute from foil suture packet and secure with 2 sutures
  7. Dress finger with bacitracin, xeroform, and 2" kling wrap
  8. Splint finger as needed with alumifoam splint (apply splint to volar side of finger so as to avoid pressure to nail bed)
  9. Repair any other lacerations as needed
  Interventions: Other: Nail Bed Repair

INTERVENTIONS:
Other: Nail Bed Repair — 1. Block involved digit with 3cc 1% lidocaine injected subcutaneously over volar and dorsal metacarpophalangeal joint
  2. Apply tourniquet to base of finger if desired
  3. Remove nail using freer/hemostats
  4. Irrigate wound with at least 500cc normal saline
  5. Repair nail bed laceration with 5-0 chromic or monocryl suture
  6. Stent eponychium with native nail or fashion substitute from foil suture packet and secure with 2 sutures
  7. Dress finger with bacitracin, xeroform, and 2" kling wrap
  8. Splint finger as needed with alumifoam splint (apply splint to volar side of finger so as to avoid pressure to nail bed)
  9. Repair any other lacerations as needed
  Arms: Nail bed repair
Other: Nail bed dressing — 1. If there is a subungual hematoma >50% of the nail, trephinate the nail plate using an 18G needle
  2. Irrigate wound with at least 500cc normal saline
  3. Dress finger with bacitracin, xeroform, and 2" kling wrap
  4. Splint finger as needed with alumifoam splint (apply splint to volar side of finger so as to avoid pressure to nail bed)
  5. Repair any other lacerations as needed
  Arms: Irrigation and Dressing

SUMMARY:
This study compares the outcomes of fixing nail bed injuries with nail bed repair versus irrigation and dressing alone. The main question this study aims to answer is "Does nail bed repair after nail bed injury lead to better outcomes?"

DETAILED DESCRIPTION:
This study compares two treatment methods for patients with nail bed injuries. The first method is irrigation and dressing. The second method is nail bed repair. Patients will be randomized into one of the two groups and outcomes will be documented in both groups.

ELIGIBILITY:
Inclusion Criteria:

* patients 2+ years of age
* presenting with disruption of nail plate or laceration adjacent to nail which appears that it may extend into the nail matrix OR subungual hematoma >50% of nail
* presenting within 3 days of acute injury

Exclusion Criteria:

* missing (e.g. avulsed) nail bed or segment of nail bed,
* prior injury to affected nail
* need for surgical treatment of injury (e.g. underlying operative fracture)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2030-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Oxford Nail Score | From time of treatment, outcomes will be measured at 1-2 weeks, 6 weeks, 1 year, and 2 years
  The Oxford Nail Score assess five cosmetic components marked as binary outcomes composed of nail shape, nail adherence, eponychial appearance, nail surface appearance and presence of a split. The final score is 0-5, where 0 is "least optimal appearance" and 5 is "most optimal appearance."

SECONDARY OUTCOMES:
Subjective Cosmesis | 1-2 weeks, 6 weeks, 1 year, 2 years
  Patients will self-score their cosmesis on a likert scale, with lower scores indicated better cosmesis. This will be scored from 0 to 8.
NRS Pain score | 1-2 weeks, 6 weeks, 1 year, 2 years
  Patients will rate their nailbed on a 0-10 scale, where 0 is no pain and 10 is the worst pain imaginable.
Nail regrowth | 1-2 weeks, 6 weeks, 1 year, 2 years
  Nail regrowth will be documented on a binary scale (yes or no) by an evaulator via photo.
Evidence of infection | 1-2 weeks, 6 weeks, 1 year, 2 years
  Evidence of infection will be evaluated on a binary scale (yes or no) by an evaluator via photo.

IPD SHARING:
Plan to Share IPD: No
We do not have plans to share this data set.

REFERENCES:
- [Background] Zook EG, Guy RJ, Russell RC. A study of nail bed injuries: causes, treatment, and prognosis. J Hand Surg Am. 1984 Mar;9(2):247-52. doi: 10.1016/s0363-5023(84)80153-7. PMID 6715836
- [Background] Ashbell TS, Kleinert HE, Putcha SM, Kutz JE. The deformed finger nail, a frequent result of failure to repair nail bed injuries. J Trauma. 1967 Mar;7(2):177-90. doi: 10.1097/00005373-196703000-00001. No abstract available. PMID 5335262
- [Background] Rao V, Akiki RK, Crozier JW, Bhatt RA, Schmidt ST, Kalliainen LK. Rethinking the Need for Nail Plate Removal: A Comparison of the Risks Between Standard Nail Bed Repair and Nonoperative Management. Ann Plast Surg. 2022 May 1;88(3 Suppl 3):S209-S213. doi: 10.1097/SAP.0000000000003197. PMID 35513322